CLINICAL TRIAL: NCT00084227
Title: A Phase Ii/Iii, Randomized, Double Blind, Comparative Trial Of Azithromycin Plus Chloroquine Versus Atovaquone-Proguanil For The Treatment Of Uncomplicated Plasmodium Falciparum Malaria In South America
Brief Title: Azithromycin Plus Chloroquine Versus Atovaquone-Proguanil For The Treatment Of Uncomplicated Plasmodium Falciparum Malaria In South America
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661126
Record Dates: First submitted 2004-06-09; First posted 2004-06-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Azithromycin; Chloroquine; atovaquone, proguanil drug combination

INTERVENTIONS:
Drug: Azithromycin/Chloroquine
Drug: Atovaquone/Proguanil

SUMMARY:
The primary objective is to confirm the hypothesis that azithromycin plus chloroquine is non-inferior to atovaquone-proguanil for the treatment of symptomatic, uncomplicated malaria due to P. falciparum.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the subject or a legally authorized representative
* Females and males >= 18 years of age with uncomplicated, symptomatic malaria as indicated by the presence of both of the following: a.) Blood smears positive for Plasmodium falciparum asexual parasitemia between 1000 - 40,000 parasites/mL; b.) Fever or history of fever (>= 38.5 C/101.2 F rectal or tympanic; >= 37.5 C/99.5 F axillary or >= 38 C/100.4 F oral) within the prior 24 hours
* Serum glucose >= 60 mg/dL (by fingerstick or peripheral blood collection)
* Positive rapid diagnostic test (Binax NOW ICT) positive for P. falciparum
* Subjects must be willing to be treated in the inpatient setting for a minimum of three days or more until parasitemia has cleared and the Investigator deems the subject fit for discharge
* Women of childbearing potential (that is, women who have not been surgically sterilized or are not clearly post-menopausal), must have a negative urine gonadotropin prior to entry into the study and must agree to use adequate contraception during the entire study and for one month after the last study visit

Exclusion Criteria:

* Severe or complicated malaria including subjects with any of the following: a.) Impaired consciousness (e.g. obtundation, unarousable coma, delirium, stupor), seizures (any seizure within a 24 hour prior to enrollment) or abnormal neurologic exam suggestive of severe or complicated malaria b.) Hemoglobinuria c.) Jaundice d.) Respiratory distress (respiratory rate â‰¥ 30 breaths/minute) e.) Persistent vomiting f.) Hematuria, as reported by the patient
* Pregnant or breast-feeding women
* History of allergy to or hypersensitivity to azithromycin or any macrolide, atovaquone, proguanil or chloroquine
* Concomitant administration of rifampin or rifabutin and metoclopramide
* History of epilepsy or psoriasis
* History of treatment with any antimalarial drug (chloroquine, quinine, mefloquine, atovaquone/proguanil, sulfadoxine/pyrimethamine, artemisinin compounds) or antibacterial with known antimalarial activity (macrolides, doxycycline, clindamycin) within 2 weeks prior to enrollment into the study
* Known or suspected cardiovascular, hepatic or renal abnormality that in the opinion of the Investigator would place the subject at increased risk to participate in the study. The following findings are specific exclusions: a.) Known or suspected creatinine clearance <30 mL/min b.) ALT and/or AST > 3 x upper limit of normal
* Inability to swallow oral medication in tablet or capsule form
* Treatment with other investigational drugs within 30 days prior to enrollment into the study
* Alcohol and/or any other drug abuse
* Requirement to use medication during the study that might interfere with the evaluation of the study drug
* Specific systemic diseases or other medical conditions that would interfere with the evaluation of the therapeutic response or safety of the study drug
* Inability to comprehend and/or unwillingness follow to the study protocol
* Prior participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2004-07; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
parasite clearance

SECONDARY OUTCOMES:
tolerability and safety

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer